CLINICAL TRIAL: NCT04575857
Title: Role of Statins In Slowing Rheumatic Heart Disease (RHD) Progression: A Feasibility Study For A Randomized Controlled Trial
Brief Title: Role of Statins In Slowing Rheumatic Heart Disease (RHD) Progression
Status: Active, not recruiting | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: Manmohan Cardiothoracic Vascular and Transplant Center (Unknown); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Nona Sotoodehnia, Co-Director, Cardiovascular Health Research Unit, University of Washington
Other Study IDs: STUDY00008837; 5R34HL143279 (NIH)
Record Dates: First submitted 2020-09-23; First posted 2020-10-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Rheumatic Heart Disease; Valvular Disease
MeSH Terms: conditions — Rheumatic Heart Disease | interventions — Atorvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Statin arm: To receive pill packet with atorvastatin (40mg/day) which will be taken nightly.
  Interventions: Drug: Atorvastatin
- Placebo arm: To receive pill packet with placebo which will be taken nightly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Participants in the intervention arm will receive a pill packet with atorvastatin (40mg) x 18 months.
  Other Names: Statin
  Groups: Statin arm
Drug: Placebo — Participants in the control arm will receive a pill packet with placebo x 18 months.
  Groups: Placebo arm

SUMMARY:
The goal of this study is to address specific implementation questions necessary and sufficient to ensure the feasibility of the larger randomized trial examining the efficacy of statin medications in slowing rheumatic heart disease (RHD) valvular pathology progression. This feasibility study is intended to confirm the number of readily recruitable subjects, assess recruitment rate, and assess the rate of valve pathology via echocardiograms. These results are necessary and sufficient to facilitate the successful design of a large full scale randomized trial to determine whether statins improve outcomes in RHD. Successful treatment of RHD would fundamentally shift the RHD management paradigm world-wide, improve the lives of millions afflicted with RHD, and subsequently, decrease health care spending on RHD management.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* History of RHD as evidenced by at least one echocardiographic examination
* No history of cardiac surgery

Exclusion Criteria:

* ≥ 75 or < 18 years old
* Absence of RHD or RF history
* Active liver disease
* Impaired hepatic and renal function, including unexplained elevated levels of alanine transaminase greater than twice the upper limit of normal
* History of previous statin intolerance or muscle disorders
* Current pregnancy (by history or lab assessment of beta hCG) or plans for pregnancy in the next 18 months). Current lactation / breast feeding.
* LDL <60

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We have developed a comprehensive electronic database of RHD/RF patients in Nepal which will serve as the main data collection and participant recruitment mechanism.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2040-02 (Estimated); Study Completion 2040-02 (Estimated)

PRIMARY OUTCOMES:
Enrollment rate | Measured at study enrollment
  Defined as the proportion of approached eligible participants who consent to enroll in the study
Medication adherence | Measured at month 1
  The investigators will conduct a pill count to assess medication adherence and will report per participant as the percent of pills taken
Medication adherence | Measured at months 6
  The investigators will conduct a pill count to assess medication adherence and will report per participant as the percent of pills taken
Medication adherence | Measured at months 12
  The investigators will conduct a pill count to assess medication adherence and will report per participant as the percent of pills taken
Medication adherence | Measured at months 18
  The investigators will conduct a pill count to assess medication adherence and will report per participant as the percent of pills taken
Retention rate | Measured at Month 18
  Proportion of enrolled participants who come for followup evaluation and remain in the study until its completion
Rate of progression of valvular disease | Change between baseline and Month 18
  Compare month 18 echocardiogram with baseline echocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Nona Sotoodehnia, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Manmohan Memorial Medical College & Teaching Hospital., Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: No